CLINICAL TRIAL: NCT02303652
Title: Surgical Treatment of Concomitant Atrial Fibrillation: a Comprehensive Insight Into Biatrial Contractility Recovery.
Brief Title: Biatrial Contractility Recovery After Maze
Status: Completed | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Claudia Loardi, MD, Centro Cardiologico Monzino
Other Study IDs: ACFA1
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Radiofrequency maze procedure — RF energy was used to create continous endocardial and epicardial lesions mimicking most of the left atrial incisions set as described in the Cox Maze III procedure. In all patients a bipolar device was used (Cardioblate BP2 Irrigated RF Surgical Ablation System®, Medtronic Inc, Minneapolis, MN, USA).
Procedure: Transthoracic echocardiography — Contemporary to clinical follow up, all patients were evaluated with 2-dimensional transthoracic echocardiography (Philips ultrasound system (iE33®, Andover, MA, USA)) at 3,6,12,24 months in order to specifically monitor the evolution of cardiac chambers dimensions and systolic performance and to record left and right atrial contractility presence.

SUMMARY:
This study aimed at evaluating multiple aspects of biatrial contractility recovery after modified maze procedure during mitral valve surgery.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a frequent complication in patients affected by mitral valve disease, causing systemic embolism, cardiac chamber dilation and decreased cardiac output. Cox et al. have designed the maze procedure as a surgical treatment for patients with AF in whom conventional therapy has failed and their lesion set is nowadays currently performed with different energy sources in order to surgically treat such supraventricular arrhythmia. In particular, the original maze was designed with three specific goals in mind: 1) the permanent AF ablation 2) the restoration of atrioventricular synchrony and 3) the preservation of atrial transport function (1). If , by one side, the efficacy of the procedure in reaching the first two goals are widely known, the restoration of the sinus rhythm does not always accompany the corresponding recovery of atrial mechanical "kick". If the atrial transport function fails to recover, benefits deriving from arrhythmia abolition might only be marginal, since, by one side, blood stasis in the atria persist, thus maintaining unchanged thromboembolic risk and, by the other side, heart hemodynamic performance is still impaired resulting from the loss of atrial contribution to cardiac output. Despite its relevant role for judging maze comprehensive success, atrial contractility outcome and clinical importance have not been deeply investigated. The purposes of this study were to evaluate by serial transthoracic echocardiography temporal modality of biatrial contractility restoration, predictive factors of atrial transport recovery and its possible relationship with cardiac chambers dimensions and function evolution after radiofrequency (RF) maze during mitral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by atrial fibrillation undergoing mitral valve surgery

Exclusion Criteria:

* Other cardiac procedures in addition to mitral valve surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by atrial fibrillation undergoing mitral valve surgery
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2005-01; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Biatrial contractility recovery after maze | 24 months
  All patients were evaluated with 2-dimensional transthoracic echocardiography at 3,6,12,24 months in order to specifically monitor the evolution of cardiac chambers dimensions and systolic performance and to record left and right atrial contractility presence.
  Transmitral flow velocity was measured with pulsed Doppler echocardiography, with a sample volume positioned at the level of the mitral tip in the apical four-chamber view and was recorded on a strip chart at a paper speed of 100 mm/s. Peak velocity and the time-velocity integral of the early filling wave (E wave) and of the late filling wave (A wave) were determined. A/E ratio, representing atrial contribution to ventricular diastolic filling, was obtained. Each measurement was obtained as an average of 6 to 8 consecutive beats.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Loardi, MD, Principal Investigator — Centro Cardiologico Monzino Milano - Italy